CLINICAL TRIAL: NCT04763083
Title: An Open-label, Phase 1, First in Human Study Investigating the Safety, Tolerability, Pharmacokinetics and Efficacy of NVG-111 in Subjects With Relapsed/Refractory ROR1+ Malignancies
Brief Title: First in Human Study of NVG-111 in Relapsed/Refractory ROR1+ Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NovalGen Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVG111-101; 2020-000820-20 (EudraCT Number)
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2022-09

CONDITIONS: Chronic Lymphocytic Leukaemia; Small Lymphocytic Lymphoma; Mantle Cell Lymphoma; Follicular Lymphoma; Diffuse Large B Cell Lymphoma; Non-small Cell Lung Cancer (NSCLC); Malignant Melanoma
Keywords: ROR1 positive cancers; Bispecific T cell engagers
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Carcinoma, Non-Small-Cell Lung; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Haematological malignancies (Experimental)
  Interventions: Drug: NVG-111
- Group B: Solid tumours (Experimental)
  Interventions: Drug: NVG-111

INTERVENTIONS:
Drug: NVG-111 — Open label, continuous iv infusion, escalating doses of NVG-111 for minimum 3 cycles

SUMMARY:
NVG-111 is a bispecific antibody drug, having two "arms", one arm attaches to a substance on cancer cells called ROR1, the other arm attaches to the body's immune cells directing them to kill the cancer cells. This is the first clinical trial of the drug NVG-111, and will include patients with certain types of cancer including chronic lymphocytic leukaemia (CLL), small lymphocytic lymphoma (SLL) mantle cell lymphoma (MCL), follicular lymphoma (FL) and diffuse large B cell lymphoma (DLBCL) in Group A. Subjects with solid tumours, focusing initially on stage IV non-small cell lung cancer (NSCLC) or malignant melanoma.

DETAILED DESCRIPTION:
Receptor tyrosine kinase-like Orphan Receptor 1 (ROR1) is a protein which is expressed at high levels on many types of cancers but is absent or expressed at low levels in normal adult organs. NVG-111 is a bispecific antibody T cell engager, comprising tandem single chain variable fragments (scFv), one arm binding to ROR1 on cancer cells, the other to cell surface CD3 on lymphocytes. Dual binding of NVG-111 causes MHC-independent immunological synapse formation, releasing perforins, granzyme B and cytokines, resulting in targeted killing of the cancer cells.

This is a Phase 1 first in human study to assess the safety, pharmacokinetics and efficacy of NVG-111 in patients with subjects with relapsed/refractory ROR1+ malignancies.

A range of doses will be studied in sequential cohorts to understand safety, pharmacokinetics and pharmacodynamics of the drug and establish the recommended phase 2 dose (RP2D). At each dose level, patients will receive 3 cycles of NVG-111 by continuous intravenous infusion, each cycle consists of 21 days treatment. Additional cycles may be given depending on the response seen.

All patients will have a safety follow up visit 4 weeks after completion of treatment with NVG-111, and will then enter long term follow up for up to two years to evaluate the duration of efficacy.

ELIGIBILITY:
Inclusion criteria:

* Personally signed informed consent document.
* Male or female, age ≥18 years.
* Relapsed or refractory ROR1+ malignancies
* ECOG performance status ≤2.
* Adequate organ function.

  * Bilirubin ≤1.5 x ULN (unless Gilbert's syndrome).
  * AST and ALT ≤2.5 x ULN (if no hepatic CLL or MCL), or AST and ALT ≤5 x ULN (if hepatic CLL or MCL).
  * APTT and PT ≤1.5 x ULN.
  * ANC ≥0.5 x 10^9 /L (without growth factors) and platelets ≥ 30 x 10^9 /L (without transfusion).
  * Serum creatinine ≤2 x ULN.
  * Estimated creatinine clearance ≥30 mL/min.
* In females of childbearing potential, a negative serum pregnancy test.
* For both males and females, willingness to use adequate contraception.
* Willingness and ability to comply with study procedures.

Exclusion Criteria:

* Richter's transformation.
* CNS or leptomeningeal active disease.
* High tumour bulk as defined in the protocol.
* Allogeneic or autologous organ transplant within prior 6 months.
* Uncontrolled autoimmune haemolytic anaemia or idiopathic thrombocytopenic purpura within 8 weeks of screening.
* Clinically significant neurological disease.
* Clinically significant cardiovascular disease or ECG abnormalities.
* Severe chronic lung disease.
* Positive test at Screening for HIV, hepatitis B or hepatitis C infection.
* Any other concurrent cancer or cancer treatments.
* Uncontrolled ongoing infection
* Recent major surgery
* Concurrent participation in another clinical trial, or experimental therapy within 5 half-lives of Screening
* Pregnant or currently breastfeeding.
* Any other medical condition that in the opinion of the investigator contraindicates participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) | Up to 10 months
  Safety parameter assessed by: type, frequency, severity and treatment-relatedness of AEs following commencement of dosing
Number of serious adverse events (SAEs) | Up to 10 months
  Safety parameter defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires inpatient hospitalisation or prolongation of existing hospitalisation, results in persistent disability/incapacity, is a congenital anomaly/birth defect, or is medically significant/important
Number of adverse events of special interest (AESI) | Up to 10 months
  Safety parameter: specific protocol-defined AEs of Grade >=3
Number of dose limiting toxicities (DLTs) | Up to 28 days
  Safety parameter assessed by protocol-defined adverse events
Laboratory safety abnormalities | Up to 10 months
  Safety parameter assessed by absolute values and change from baseline in laboratory safety assessments
Vital sign abnormalities | Up to 10 months
  Safety parameter assessed by absolute values and change from baseline in vital signs
ECG abnormalities | Up to 10 months
  Safety parameter assessed by absolute value and change from baseline in ECG intervals including QTcF
Changes from baseline in ECOG | Up to 10 months
  Safety parameter assessed by change from baseline in ECOG performance status

CONTACTS AND LOCATIONS:
Overall Officials: Parag Jasani, MBBS, FRCP, FRCPath, Principal Investigator — Royal Free London NHS Foundation Trust and University College London Hospitals
Locations (3):
- United Kingdom (3):
  - University College London Hospital, London
  - Royal Marsden Hospital, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Undecided
The company is developing an IPD sharing plan which will be completed and posted prior to primary completion date of the study